CLINICAL TRIAL: NCT00561392
Title: A 24-week, Multi-center, Open, Evaluation of the Clinical Effectiveness of the Once-daily 10 cm^2 Rivastigmine Patch Formulation in Patients With Probable Alzheimer's Disease (MMSE10-26)
Brief Title: Clinical Effectiveness of 10 cm^2 Rivastigmine Patch in Patients With Alzheimer's Disease
Acronym: ADEPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CENA713DDE15
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Rivastigmine; Patch
MeSH Terms: conditions — Alzheimer Disease

ARMS (1):
- Rivastigmine 5 and 10 cm^2 patch (Experimental): For the 1st 4 weeks of this 24 week study, patients were administered rivastigmine transdermally once daily via a 5 cm^2 patch. After the Week 4 assessment, patients were administered rivastigmine transdermally once daily via a 10 cm^2 patch, with adjustments as necessary for safety and tolerability.
  Interventions: Drug: Rivastigmine 5 and 10 cm^2 patch

INTERVENTIONS:
Drug: Rivastigmine 5 and 10 cm^2 patch

SUMMARY:
This study evaluated the safety and efficacy of 10 cm^2 rivastigmine patch in patients with Alzheimer Disease (MMSE 10-26). The primary objective was the percentage of patients who stayed on the target size of 10 cm^2 for at least 8 weeks. This proportion was then compared to historical data of the percentage of patients who could reach a rivastigmine capsule target dose of 12 mg and stay on it at least 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males, and females not of child-bearing potential (surgically sterile or at least one year postmenopausal), of at least 50 years of age
* Probable Alzheimer's disease according to the NINCDS-ADRDA (National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association) and DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) criteria
* MMSE (Mini-Mental State Examination) score of > 10 and < 26
* Patients initiating therapy for the first time with a cholinesterase inhibitor (patients prescribed both rivastigmine and memantine are allowed)
* Patients who failed to benefit from previous cholinesterase inhibitor treatment

Exclusion Criteria:

* Patients not treated according to the product monograph for rivastigmine capsules
* patients involved in a clinical trial
* Current diagnosis of an active skin lesion/disorder that would prevent accurate assessment of the adhesion and potential skin irritation of the patch (e.g., atopic dermatitis, wounded or scratched skin in the area of the patch application)

Other protocol-defined exclusion criteria applied to the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Munich, Germany

REFERENCES:
- [Derived] Articus K, Baier M, Tracik F, Kuhn F, Preuss UW, Kurz A. A 24-week, multicentre, open evaluation of the clinical effectiveness of the rivastigmine patch in patients with probable Alzheimer's disease. Int J Clin Pract. 2011 Jul;65(7):790-6. doi: 10.1111/j.1742-1241.2011.02713.x. Epub 2011 Jun 6. PMID 21645184

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Started | 208
Completed | 155
Not Completed | 53
Not completed — Adverse Event | 38
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 8
Not completed — Administrative problems | 4

BASELINE CHARACTERISTICS:
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 208
Age Continuous [Mean (Standard Deviation); unit: years] | 74 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 98
Region of Enrollment [Number; unit: participants]
  Germany | 208

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Treated by Rivastigmine 10 cm^2 Patch for at Least 8 Weeks Who Completed the Study
Description: Dosages of study medication prescribed to and taken by the patient was assessed in a "Drug Administration Record" with start date, end date, dosage and reason for dose adjustment (if applicable). Data was amended by counting the returned medication at the study visits and information by the caregiver.
Time Frame: Baseline to Week 24
Population: The Intent-to-Treat (ITT) population was defined as all randomized patients who were administered at least one dose of study medication and were assessed at baseline and post-baseline for efficacy at least 1 time.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 182
Percentage of participants | 74.2 [67.8 to 80.5]

2. Secondary Outcome: Mean Change From Baseline in the Mini-Mental State Examination (MMSE) Score at Week 24
Description: The MMSE is a brief, practical screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 182
Units on a scale | 1.3 (3.8)

3. Secondary Outcome: Mean Change From Baseline in the Trail-making Test Part A Score at Week 24
Description: The Trail-making test is a neuropsychological test of visual attention and task switching. The task requires a subject to 'connect-the-dots' of 25 consecutive numbers (1,2,3, etc.) on a sheet of paper or computer screen. The goal of the subject is to finish the test as quickly as possible, and the time taken to complete the test is used as the primary performance metric (in seconds). The maximum time allowed is 300 seconds. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 182
Seconds | -8.9 (109.45)

4. Secondary Outcome: Mean Change From Baseline in the Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) Score at Week 24
Description: The ADCS-ADL scale is composed of 23 items developed to assess a patient's performance of both basic and instrumental activities of daily living such as those necessary for personal care, communicating and interacting with other people, maintaining a household, conducting hobbies and interests, as well as making judgments and decisions. Responses for each item will be obtained from the caregiver through an interview. The range for the total ADCS-ADL score is 0 to 78; a higher score indicates a more self-sufficient individual. A positive change score indicates improvement.
Time Frame: Baseline to Week 24
Population: The Intent-to-Treat (ITT) population was defined as all patients who were administered at least one dose of study medication and were assessed for efficacy at least 1 time.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 182
Units on a scale | 1.3 (12.02)

5. Secondary Outcome: Change From Baseline in the Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change (ADCS-CGIC) at Week 24 Assessed by the Physician
Description: The ADCS-CGIC is an assessment tool to make a judgment of change in a patient's condition. Change is derived from comparing an assessment performed at baseline versus an assessment at the end of the study. Change is categorized into 1 of 7 categories: No change; minimal, moderate, or marked improvement; or minimal, moderate, or marked decline. Results are reported as number of patients in the indicated change category.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 182
Participants
  No change | 47
  Minimal improvement | 25
  Moderate improvement | 23
  Marked improvement | 15
  Minimal decline | 37
  Moderate decline | 12
  Marked decline | 5

6. Secondary Outcome: Mean Change From Baseline in the Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change (ADCS-CGIC) at Week 24 Assessed by the Caregiver
Description: The ADCS-CGIC is an assessment tool to make a judgment of change in a patient's condition. Change is derived from comparing an assessment performed at baseline versus an assessment at the end of the study. Change is categorized into 1 of 7 categories: No change; minimal, moderate, or marked improvement; or minimal, moderate, or marked decline.
Time Frame: Baseline t0 Week 24
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 182
Participants
  No change | 21
  Minimal improvement | 23
  Moderate improvement | 16
  Marked improvement | 15
  Minimal decline | 56
  Moderate decline | 20
  Marked decline | 14

7. Primary Outcome: Percentage of Participants Treated by Rivastigmine 10 cm^2 Patch for at Least 8 Weeks Regardless Whether They Completed the Study
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 182
Percentage of participants | 80.8 [75.0 to 86.5]

8. Primary Outcome: Percentage of Participants Who Were Compliant to the 10 cm^2 Patch
Description: as for outcome 1
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 182
Percentage of participants | 95.0 (28.3)

9. Secondary Outcome: Mean Change From Baseline in the Mini-Zarit Inventory Score of Caregiver Burden at Week 24
Description: The Mini-Zarit Inventory assesses the burden of a caregiver in caring for a patient. The inventory is composed of 5 questions which are rated according to the following answers: 0 = never, ½ = sometimes, 1 = often. The ratings on the 5 questions are added together resulting in a total score of 0 to 7 with a higher score indicating greater caregiver burden. A negative change score indicates reduced burden.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Number analyzed (Participants) | 182
Units on a scale | 0.4 (1.58)

ADVERSE EVENTS:
Arm/Group | Rivastigmine 5 and 10 cm^2 Patch
Serious Adverse Events (participants affected / at risk) | 18/208
Other Adverse Events (participants affected / at risk) | 49/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine 5 and 10 cm^2 Patch (N=208)
Bradycardia (Cardiac disorders) | 1
Death (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Blood glucose abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 3
Dysstasis (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Aggression (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 2
Disorientation (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivastigmine 5 and 10 cm^2 Patch (N=208)
Nausea (Gastrointestinal disorders) | 21
Vomiting (Gastrointestinal disorders) | 15
Erythema (Skin and subcutaneous tissue disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.